CLINICAL TRIAL: NCT04831606
Title: A Single-center Prospective Randomized Controlled Study on the Efficacy of Blue Light in the Therapy of Neuro-ischemic Foot Lesions in Patients With Type I or II Diabetes in a Combined Hospital /Territory Treatment Regimen.
Brief Title: Blue Light Photobiomodulation Therapy on Neuroischemic Patients
Acronym: HERMES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: very low enrollment rate
Sponsor: Emoled (Industry)
Collaborators: Ospedale San Donato (Other); University of Pisa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EmoLED_DF_001
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Debridement

STUDY DESIGN:
Intervention Model Description: A double-blind pilot trial on outpatients affected by diabetic foot ulcers, followed in an integrated way by both a specialized center and the home nursing network, for a period of 24 weeks.
  The specialist center will characterize the patient, set the therapy, and evaluate them monthly, the nursing service will treat them at home biweekly.
  The physician in charge of the monthly evaluation is unaware of the patient's arm. During therapy, the patient will wear blinding glasses, the control arm will simulate the use of the device switching it on without aiming it at the wound.
  After a two-week pre-enrollment period to evaluate the wound progression applying only the standard care (if the wound reduces 50% or more, the patient will be excluded), the patient will be randomized into one of the study arms: the control arm will continue with the standard treatment, while the EmoLED Arm will receive EmoLED's therapy in addition to the standard treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized into the two arms of the study according to a list of random numbers generated by special IT tools and communicated by the scientific supervisor to the Care Provider via e-mail .
  It is a 1: 1, single-block randomization of 40 patients distributed in the two groups (treated and control). After the two-week enrollment observation period, the Investigator at the outpatient center will ascertains the conditions for the study prosecution and will notify the Head of the Care Providers to take charge of the patient included in the study and to proceed with the assignment to one of the groups. In this way, the Investigator at the outpatient center will be blinded to the treatment performed at home by the patient.
  All patients will receive a pair of blinding glasses at the enrollment and will be required to wear them during therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Patients will receive a biweekly standard treatment at home according to the International Working Group on Diabetic Foot consisting of: Debridement of the lesion, unloading with a brace up to the calf, non-removable (except for contraindications), dressing of the wound with advanced dressings in use at the specialized center and in the home care network.
  Interventions: Procedure: debridement; Device: Offloading; Device: Advanced dressing
- EmoLED Arm (Experimental): Patients on top of the standard treatment of the control arm will receive EmoLED blue light irradiation for two minutes at each biweekly medication.
  Interventions: Procedure: debridement; Device: Offloading; Device: Advanced dressing; Device: Blue Light Photobiomodulation

INTERVENTIONS:
Procedure: debridement — Cleaning of the wound area
Device: Offloading — Offloading performed with a standard brace to the calf (Optima Diab, from Molliter).
Device: Advanced dressing — Protect the wound with Advanced dressing
Device: Blue Light Photobiomodulation — 2 minutes irradiation of blue light performed with EmoLED device
  Arms: EmoLED Arm

SUMMARY:
This is a pilot case/control clinical study on a group of outpatients with diabetic foot lesions aiming to verify the efficacy and safety of the Blue light photobiomodulation therapy with EmoLED medical device, in addition to standard therapy compared to the standard therapy alone, evaluating the percentage of healed lesions (which have reached complete and lasting re-epithelialization), the evaluation of the healing time and reduction of the ulcerated area during the time of observation, the perception of pain and the quality of life of the enrolled patients.

The aim of this study is therefore to determine any differences in outcome between the two groups considered and, in particular, if the therapy of the group being treated is more effective than the standard therapy in terms of percentage of healed lesions, healing time, and reduction of the ulcerated area, pain perception, and quality of life, and is at least as safe in terms of occurrence of adverse events.

DETAILED DESCRIPTION:
This study will be conducted according to the standards of Good Clinical Practice and in compliance with the principles set out in the Declaration of Helsinki, with the UNI_ISO_14155_2011 standard, and with all relevant local laws and regulations applicable to clinical trials that use patients as the research object. This clinical investigation in the various centers involved cannot begin before having received the favorable written approval of the Ethics Committee of the coordinating center and the respective Ethics Committees. The medical assistance provided to the subject is the responsibility of adequately qualified doctors, as all the centers involved in this study are centers specialized in the treatment of the pathology object of the clinical trial (Diabetology units or Diabetic Foot clinics).

During this trial, the patients' right to physical and mental integrity, the right to privacy, and the protection of data concerning them will be respected following Directive 95/46/EC.

This clinical investigation has been designed in such a way as to cause as little pain, discomfort, fear, and other foreseeable risks for the subject as possible and the degree of discomfort related to the trial itself or the treatment with the medical device in question is almost nil, considered the clinical evaluation report of the device and the safety data obtained from post-marketing surveillance.

The degree of discomfort/pain of the enrolled patients is however subject to continuous verification during the clinical trial, through a special questionnaire on the detection of discomfort connected to participation in the study in question. The risk/benefit ratio will be constantly checked throughout the trial, taking into account any adverse events / device-related accidents or non-serious side effects reported by the main investigators, and the preliminary assessment of the benefits found on patients who have completed the study process.

The principal investigator of each center is responsible for adequate conduct of the study of his own center and the coordination of the personnel involved. Must be responsible for all medical decisions relating to the study and ensure that adequate medical assistance is provided to the subject in case of adverse events. The investigator should conduct the study following the protocol agreed with the sponsor and the authorities.

To verify that the rights, safety, and well-being of enrolled patients are protected, that the data communicated are reliable and solid, and that the clinical investigation is conducted in compliance with the prescriptions of current legislation, the sponsor guarantees adequate monitoring of the conduct of this clinical investigation. The monitoring of the clinical investigation is entrusted to the sponsor's staff adequately trained. To ensure compliance with ICH/GCP guidelines and current legislation, such personnel will be responsible for ensuring that the Study is conducted in full compliance with the Standard Operating Procedures, the Protocol, and other written instructions.

The main responsibilities of the personnel carrying out the monitoring are to ensure adherence to the Protocol, to ensure that data is recorded and reported accurately and completely, and to verify that informed consent has been obtained and recorded for all subjects before they participate in the study. Researchers will be contacted at regular intervals throughout the study period. To check and verify the various documents (Data Collection Cards or CRFs and other relevant documents containing the original data) relating to the Study to verify compliance with the Protocol and to ensure the completeness, consistency, and accuracy of the recorded data.

Monitoring staff will conduct a center opening visit (SIV), a minimum of three visits during the study (MOV) to be scheduled approximately one after 1 or 2 months after SIV based on the number of patients enrolled, one at two-thirds of the enrollment and another after the observations on the last patient. Finally, once all the open issues have been resolved (open queries, clarifications, etc.), we will proceed with the center closing visit (COV). Should additional monitoring visits be necessary, the staff will schedule them with the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from neuro-ischemic diabetic foot ulcer grade IC or IIC according to the University of Texas Wound Classification; If the patient has two or more lesions, which may fall within the inclusion criteria, the most serious lesion (index lesion) will be selected and followed for the entire duration of the study.
* Patients who, following hospital discharge or after the first outpatient assessments, are followed by Home Care and are always monitored at the same referral center;
* Patients with type I or II diabetes, with blood glucose ≤ 10%;
* Patients willing to constantly wear the offload braces prescribed by the reference center;
* Patients with ulcer localized on the finger, lateral, plantar, or dorsal part of the foot with an extension greater than 1 sqcm;
* Patients with confirmed neuropathy with Monofilament (Semmes-Weinstein 5.07 / 10g);
* Patients with ABPI between 0.7 - 0.9, ankle PA> 70mmHg, TcPO2 between 36 - 50 mmHg;
* Patients with lesions lasting between 1 and 24 months;
* Patients who understand the purpose of the Clinical Study and provide their informed consent in writing.

Exclusion Criteria:

* Patients who have participated in a clinical study with a drug or medical device for less than a month;
* Patients who are unable to understand the aims and objectives of the study;
* Patients who are bedridden or unable to walk or Patients with neoplasms;
* Patients with pressure ulcers;
* Patients who have infectious signs according to IDSA criteria;
* Patients who underwent revascularization in the previous two months;
* Patients who have presented an acute ischemic event within the previous 3 months;
* Patients with heel injuries;
* Patients with nephropathy undergoing dialysis;
* Patients with osteomyelitis;
* Patients with Charcot's neuro-arthropathy:
* Patient on high dose corticosteroid therapy (≥ 40 mg/day);
* Patients with a history of self-harm who can voluntarily alter the course of healing;
* Patients with psychiatric disorders;
* Women who are pregnant or breastfeeding;
* Patients with pathologies or under treatment with drugs that induce photosensitization of the skin;
* Patients with a life expectancy of less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Percentage of healed lesions on the total lesions treated for each arm | 24 weeks (20 weeks treatment plus 4 weeks post treatment observation)
  Percentage of lesions showing a lasting and complete re-epithelialization in each group after twenty-four weeks.
  Healing must be confirmed by the Principal Investigator or his staff during an outpatient visit at the reference center participating in the study

SECONDARY OUTCOMES:
Healing time | 24 weeks
  Number of days needed to reach a lasting and complete re-epithelialization within the observation period

OTHER OUTCOMES:
Reduction of the lesion surface in both arms, measured in absolute terms (square centimeters) and as % of the initial size. | once every 4 weeks for 20 weeks plus the last control visit at 24 weeks if needed
  At each outpatient control visit, a photograph image will be acquired with the device in the use of the structure (WoundViewer from Omnidermal Biomedics Srl). The device takes pictures and calculates automatically the area of the wounds through a validated algorithm.
Quality of life level (QoL), measured with specific questionnaires (EuroQoL-5D) | 16 weeks (last outpatient visit)
  At the first and last visit in the outpatient center information on the patient's quality of life will be collected using standard models such as the EQ-5D and the Wound-QoL both available and validate in the Italian language.
Pain perception measured according to the VAS scale | 20 weeks
  At each visit the patient pain perception will be measured using the standard VAS scale method
Comparative Evaluation of costs associated with the therapy. | 16 weeks
  Both sanitary costs and patients' costs (including caregiver if present) in connection with the therapy will be recorded. Through a questionnaire to be filled at the last visit by the patient, the caregiver, the home nurse, and the outpatient center all direct, indirect, medical personnel, and societal costs will be recorded.
  the home nurses and outpatient center will fill a questionnaire regarding direct and indirect costs connected with the therapy for both arms.
Patient's therapy acceptance | 24 weeks
  at the control visit a questionnaire to evaluate the therapy's acceptance will be given to patients of both arms.
Appreciation, complexity and usefulness of the EmoLED therapy by the operator | 24 weeks
  a specific questionnaire will be administered to the personnel to evaluate appreciation, complexity and usefulness of the EmoLED therapy.
Number of Treatment-Emergent Adverse Events | 24 weeks
  All incidents according to the definition of the EU regulation 2017/745 on Medical Devices will be properly reported their gravity and relation with the therapy evaluated.
  It will be counted the number and gravity of occurred adverse events on both arms
Evaluation of cost-effectiveness of using EmoLED for the treatment of ulcers | 24 weeks
  Evaluation of cost-effectiveness using EmoLED in the treatment of ulcers through economic-organizational impact survey.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Piaggesi, Doctor, Study Chair — Pisa University Hospital; Alessia Scatena, Doctor, Principal Investigator — San Donato Hospital
Locations (1):
- San Donato Hospital, Arezzo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenhalgh DG. Management of Burns. N Engl J Med. 2019 Jun 13;380(24):2349-2359. doi: 10.1056/NEJMra1807442. No abstract available. PMID 31189038
- [Background] Mast BA, Schultz GS. Interactions of cytokines, growth factors, and proteases in acute and chronic wounds. Wound Repair Regen. 1996 Oct;4(4):411-20. doi: 10.1046/j.1524-475X.1996.40404.x. PMID 17309691

DOCUMENTS (1):
  • Study Protocol (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT04831606/Prot_001.pdf